CLINICAL TRIAL: NCT03906825
Title: Acute Effects of Curcuminoids, EPA (Omega-3), Astaxanthin and GLA (CEAG) on Inflammation and Endothelial Function
Brief Title: Effect of CEAG on Inflammation and Endothelial Function
Acronym: CEAG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Responsible Party: Principal Investigator, Matthew J. Budoff, M.D;FACC, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 22051-01
Record Dates: First submitted 2019-03-29; First posted 2019-04-08 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Inflammation; Endothelial Dysfunction
Keywords: Endothelium
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: Double Blind Placebo Controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dietary supplement CEAG (Active Comparator): The dietary supplements consists of Curcuminoids, EPA (Omega-3), Astaxanthin and GLA (CEAG).
  Interventions: Dietary Supplement: CEAG
- Placebo (Placebo Comparator): The Placebo does not contain any CEAG.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: CEAG — Curcuminoids, EPA (OMEGA-3), Astaxanthin, GLA
  Arms: dietary supplement CEAG
Dietary Supplement: placebo — placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to look at the effect a dietary supplement called CEAG [Curcuminoids, EPA (Omega-3), Astaxanthin and Gamma Linolenic Acid (GLA)] has on inflammation and endothelial (inner layer of the blood vessels) function and whether it causes a lowering of blood pressure.The endothelium plays in an important role in blood pressure.

DETAILED DESCRIPTION:
This clinical trial is to assess the efficacy of Curcuminoids, EPA (Omega-3), Astaxanthin and GLA for improving inflammation and endothelial reactivity over a four week intervention period in individuals with metabolic syndrome. The study also examines the effect of Curcuminoids, EPA (Omega-3), Astaxanthin and GLA administration on other markers of cardiovascular function and cardiovascular disease risk including Total, LDL and HDL-Cholesterol, Triglycerides, and a multitude of inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* age 18-75 years
* BP 121-140/81-90 mm Hg on average
* Body Mass Index (BMI) 18-40.

Exclusion Criteria:

* free of chronic diseases including cancer or rheumatologic disorders
* weight in excess of 350 pounds
* bleeding disorder
* history of myocardial infarction or all types of revascularization procedures, second or third degree heart block with or without a pacemaker
* angina pectoris of any type
* concurrent potentially life-threatening arrhythmia or symptomatic arrhythmia clinically significant valvular heart disease
* history of malignancy of any organ system, treated or untreated, within the past 5 years whether or not there is evidence of local recurrence or metastases, (with the exception of localized basal cell carcinoma of the skin)
* serum creatinine > 2.0 mg/dl
* concurrent enrollment in another placebo-controlled trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2018-08-13 (Actual); Study Completion 2018-08-13 (Actual)

PRIMARY OUTCOMES:
change from baseline in inflammation at 4 weeks | 4 weeks
  Inflammatory markers IL-6, CRP

SECONDARY OUTCOMES:
Rate of change from baseline of endothelial function | 4 weeks
  endothelial function measured by brachial artery flow mediated dilatation
Rate of change in cardio-metabolic relevant biomarkers | 4 weeks
  Cardio-metabolic relevant biomarkers including fasting Lipids (mg/dL), Glucose (mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Budoff, MD, Principal Investigator — Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Locations (1):
- Lundquist Institute for Biomedical Innovation at Harbor UCLA Medical Center, Torrance, California, United States

REFERENCES:
- [Derived] Birudaraju D, Cherukuri L, Kinninger A, Chaganti BT, Shaikh K, Hamal S, Flores F, Roy SK, Budoff MJ. A combined effect of Cavacurcumin, Eicosapentaenoic acid (Omega-3s), Astaxanthin and Gamma -linoleic acid (Omega-6) (CEAG) in healthy volunteers- a randomized, double-blind, placebo-controlled study. Clin Nutr ESPEN. 2020 Feb;35:174-179. doi: 10.1016/j.clnesp.2019.09.011. Epub 2019 Oct 24. PMID 31987113